CLINICAL TRIAL: NCT00668655
Title: An Evaluation of the Cosmetic Appearance of Metronidazole Gel (MetroGel®) 1%
Status: Completed | Type: Observational
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Other Study IDs: US10086
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2012-09

CONDITIONS: Rosacea
Keywords: Rosacea, metronidazole
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Female Subjects aged 20 to 75 inclusive, with a diagnosis of moderate (Global Severity Score of 3) Rosacea
  Interventions: Drug: Metronidazole Gel

INTERVENTIONS:
Drug: Metronidazole Gel — Topical, Once daily for 2 weeks
  Other Names: MetroGel® 1%

SUMMARY:
The purpose of this study is to determine the cosmetic appearance of metronidazole gel (MetroGel®) 1% with commonly marketed facial foundations.

DETAILED DESCRIPTION:
Evaluate the relationship between treatment with MetroGel® 1% and cosmetic performance with the Subjects' usual cosmetic products. It is expected that the female subjects will be able to use their routine cosmetics after application without affecting the cosmetic product's performance or causing side effects.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate Rosacea (Global Severity Score of 3),
* Subjects willing to stop their current rosacea medication for at least 2 weeks
* Subjects must have an established routine of cosmetics application (e.g. must have been using the same facial foundation for at least 3 months and it is not expected to change during the study)
* Subjects must be willing to use their routine facial foundation and not change products while on study

Exclusion Criteria:

* Subjects who do not routinely wear facial foundation
* Subjects who failed to undergo a washout period of 14 days for the use of topical rosacea therapy, (for example: metronidazole, azelaic acid, sulfacetamide)
* Subjects who are unwilling to stop their current rosacea medications for 2 weeks

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

SECONDARY OUTCOMES:
Assessment of Cosmetic Appearance by Investigator | Baseline and Week 2
Assessment of Cosmetic Appearance by Subject | Baseline and Week 2
Erythema Severity | Baseline and Week 2
Investigator Global Severity Score | Baseline and Week 2
Tolerability Assessments and incidence of adverse events | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ronald W Gottschalk, MD, Study Director — Galderma R&D
Locations (1):
- Dermatology Consulting Services, High Point, North Carolina, United States

REFERENCES:
- [Derived] Draelos ZD, Colon LE, Preston N, Johnson LA, Gottschalk RW. The appearance of facial foundation cosmetics applied after metronidazole gel 1%. Cutis. 2011 May;87(5):251-9. PMID 21699130